CLINICAL TRIAL: NCT01832818
Title: A Prospective, Feasibility, Multi-Center Nonrandomized Clinical Trial Evaluating the Safety and Effectiveness of NuNec® Cervical Arthroplasty System
Brief Title: Post-Market Study Evaluating the Safety and Effectiveness of NuNec® Cervical Arthroplasty System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has been terminated early due to slow enrolment.
Sponsor: Pioneer Surgical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C01
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Cervical Intervertebral Disc Degeneration
Keywords: Total Disc Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NuNec Cervical Disc (Experimental): Each patient will be implanted with the NuNec Cervical Disc in a single level from C3 to C7. Postoperatively, patient evaluated at discharge, 6 weeks, 3, 6, 12 and 24 months.
  Interventions: Device: NuNec Cervical Disc

INTERVENTIONS:
Device: NuNec Cervical Disc — Patients will be enrolled and implanted with the NuNec device at a single level C3 to C7.
  Other Names: NuNec Cervical Arthroplasty System

SUMMARY:
The objective of this study is to evaluate long-term safety and effectiveness of the NuNec® Cervical Arthroplasty System in a small patient population. The NuNec device is currently CE marked and commercially available in Europe.

DETAILED DESCRIPTION:
The NuNec® feasibility study is a prospective, multi-centered, non-randomized clinical trial. Only patients who have been diagnosed with single level, C3 to C7, symptomatic cervical degenerative disc disease and have failed at least 6 weeks of conservative treatment or present signs of progression of spinal cord/nerve root compression with continued non-operative care will be enrolled.

Patients will be evaluated preoperatively and postoperatively at discharge, 6 weeks, 3, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* is at least 21 years of age and skeletally mature
* must have symptomatic degenerative disc disease at one level in the cervical spine, C3 to C7, demonstrated by herniated disc and/or spondylosis;
* must have completed a minimum of six weeks of unsuccessful conservative, non-operative care or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of conservative treatment
* must score at least 15/50 (30%) on the Neck Disability Index
* is willing and able to follow the post-operative management program
* must understand and sign the informed consent document

Exclusion Criteria:

* symptomatic cervical DDD at more than one level
* axial neck pain as the primary diagnosis without evidence of neural compression
* neck or arm pain of unknown etiology
* any significant anatomical consideration which would make the anterior cervical approach excessively risky or impossible
* severe spondylosis at the target level
* prior surgery at the target level
* fused level adjacent to the target level
* osteoporosis, osteopenia, osteomalacia, Paget's disease or metabolic bone disease
* active infection or surgical site infection
* is using any medication known to interfere with bone/soft tissue healing
* diabetes mellitus requiring daily insulin management
* any terminal, systemic, or autoimmune disease
* medical conditions or mental incompetence which may interfere with study requirements
* BMI >40 or a weight more than 100 lbs over ideal body weight
* chemical dependency problem that may interfere with study requirements
* current smokers
* history of any invasive malignancy unless treated and in remission for at least two years
* documented allergies to metal or plastic
* currently pregnant, or interested in becoming pregnant during the study follow-up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tai Friesem, MD, Principal Investigator — University Hospital of North Tees
Locations (1):
- University Hospital of North Tees, Stockton-on-Tees, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NuNec Cervical Disc
Started | 14
Completed | 8
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | NuNec Cervical Disc
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Neck Disability Index (NDI) Score Improvement of at Least 15 Points
Description: The Neck Disability Index is a patient reported outcome measure for self-rated disability due to neck pain. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score. A higher score would indicate that the patient did not improve.
Time Frame: At 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NuNec Cervical Disc
Number analyzed (Participants) | 8
units on a scale | 28.4 (27.1)
Statistical Analysis 1: Comparison: NuNec Cervical Disc; Test type: Superiority; p < 0.05, ANOVA

2. Primary Outcome: Visual Analog Scale (VAS) Improvement of 2.0 cm for Neck Pain
Description: The pain Visual Analog Scale is a uni-dimensional measure of pain intensity, represented by a 100 mm line, anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]). A higher score would indicate that the patient had a worse outcome.
Time Frame: At 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NuNec Cervical Disc
Number analyzed (Participants) | 8
units on a scale | 2.97 (3.27)
Statistical Analysis 1: Comparison: NuNec Cervical Disc; Test type: Superiority; p < 0.05, ANOVA

3. Primary Outcome: Serious Adverse Events Related to the Device
Description: The number of serious adverse events have been recorded
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | NuNec Cervical Disc
Number analyzed (Participants) | 8
Participants | 0

4. Primary Outcome: Device Failures or Removals, Revisions, Re-operations
Description: The failures or re-operations or supplemental fixation at the treated level
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | NuNec Cervical Disc
Number analyzed (Participants) | 8
Participants | 0

5. Secondary Outcome: Patient Satisfaction
Description: As assessed on patient questionnaire.
Time Frame: At 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | NuNec Cervical Disc
Number analyzed (Participants) | 8
Participants
  Very Satisfied | 3
  Satisfied | 4
  Somewhat Satisfied | 1
  Unsatisfied | 0

6. Secondary Outcome: Absence of Device Migration or Subsidence
Description: Absence of device migration > 3mm; Absence of device subsidence > 3mm
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | NuNec Cervical Disc
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over the 24 month follow-up period
Arm/Group | NuNec Cervical Disc
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NuNec Cervical Disc (N=14)
neurological impairment (Nervous system disorders) | 1 (1) — 1 patient developed a neurological impairment, this was not considered related to the surgery or the device.
Dysphagia (Musculoskeletal and connective tissue disorders) | 1 (1) — Ongoing Dysphagia (mainly to solids), hoarse voice ( improving)
Pain in L forearm (Musculoskeletal and connective tissue disorders) | 1 (1)
Hand Paranesthesia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperesthesia (Musculoskeletal and connective tissue disorders) | 1 (1) — Hyperesthesia C5/6 distribution L arm
Limited shoulder movement (Musculoskeletal and connective tissue disorders) | 1 (1) — Limited movement L shoulder

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No